CLINICAL TRIAL: NCT05131178
Title: Double Blind Randomized Trial of Post-operative Cesarean Continuous Infusion of Bupivacaine Versus Placebo for Local Incisional Pain Control
Brief Title: Post-operative Cesarean Trial of Pain Control
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Avanos Medical (Other); Children's Hospital Colorado (Other); Colorado Fetal Care Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 21-2810
Record Dates: First submitted 2021-11-10; First posted 2021-11-23 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Post-operative Pain; Cesarean Section
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Saline (Placebo Comparator): ON-Q Pump® with continuous infusion of saline (270 mL of normal saline)
  Interventions: Device: ON-Q Pump® with continuous infusion of saline
- Bupivacaine (Experimental): ON-Q Pump® with continuous infusion of bupivacaine (270 ml of 0.5 % bupivacaine)
  Interventions: Device: ON-Q Pump® with continuous infusion of bupivacaine

INTERVENTIONS:
Device: ON-Q Pump® with continuous infusion of bupivacaine — 270 ml of 0.5 % bupivacaine. The device being used is a fixed flow pump meaning the rate of 2 mL/hour. The pump is connected to the catheter and left in place for up to 4 post-operative days or until the completion of the infusion.
  Arms: Bupivacaine
Device: ON-Q Pump® with continuous infusion of saline — 270 mL of normal saline. The device being used is a fixed flow pump meaning the rate of 2 mL/hour. The pump is connected to the catheter and left in place for up to 4 post-operative days or until the completion of the infusion.
  Arms: Saline

SUMMARY:
This study plans to learn more about postoperative pain management after cesarean deliveries (C-sections). As a part of standard of care, the Children's Hospital Colorado's Colorado Fetal Care Center (CFCC) follows the standard Enhanced Recovery After Cesarean (ERAC) guidelines to manage pain following C-section delivery. In addition, the CFCC uses an FDA approved medical device called the ON-Q ® Pump, which continuously delivers local anesthetic medication to control pain in the area of your procedure. The local anesthetic used is bupivacaine, which is FDA approved for use to control local pain after C-sections. The CFCC has found a significant reduction in opioid use after adopting both of these procedures. The study aims to determine if the ERAC protocol or ON-Q ® Pump continuous infusion is responsible for lower opioid use by comparing bupivacaine (treatment) versus saline (placebo) groups.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients 18 years of age or older
* Patients undergoing both scheduled and unscheduled cesarean deliveries at CFCC

Exclusion Criteria:

* Active substance abuse (ex methamphetamines) determined by patient report, toxin screen, or screening physician's determination
* Current treatment for chronic pain involving opiate receptor agonism or antagonism (i.e. suboxone, methadone, naltrexone, oxycodone)
* Contraindication to neuraxial anesthesia
* Known allergies to common anesthetic medications
* Inability to consent to study procedures
* Patient receiving general anesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-11-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Total postoperative opioid use | Post-operative day 4
  Total postoperative opioid use in morphine equivalents through discharge

SECONDARY OUTCOMES:
Patient satisfaction survey with Visual Analog Scale (VAS) Pain Score | At hospital discharge (about post-operative day 5)
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (score of 0) and "worst pain" (score of 100 [100-mm scale]).
Antiemetic use at Baseline | Baseline
  Daily antiemetic use by number of doses through discharge
Antiemetic use at post-operative day 1 | Post-operative day 1
  Daily antiemetic use by number of doses through discharge
Antiemetic use at post-operative day 2 | Post-operative day 2
  Daily antiemetic use by number of doses through discharge
Antiemetic use at post-operative day 3 | Post-operative day 3
  Daily antiemetic use by number of doses through discharge
Antiemetic use at post-operative day 4 | Post-operative day 4
  Daily antiemetic use by number of doses through discharge
Antiemetic use at hospital discharge (about post-operative day 5) | At hospital discharge (about post-operative day 5)
  Daily antiemetic use by number of doses through discharge
Visual Analog Scale (VAS) Pain Score at Baseline | Baseline
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (score of 0) and "worst pain" (score of 100 [100-mm scale]).
Visual Analog Scale (VAS) Pain Score at post-operative day 1 | Post-operative day 1
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (score of 0) and "worst pain" (score of 100 [100-mm scale]).
Visual Analog Scale (VAS) Pain Score at post-operative day 2 | Post-operative day 2
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (score of 0) and "worst pain" (score of 100 [100-mm scale]).
Visual Analog Scale (VAS) Pain Score at post-operative day 3 | Post-operative day 3
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (score of 0) and "worst pain" (score of 100 [100-mm scale]).
Visual Analog Scale (VAS) Pain Score at post-operative day 4 | Post-operative day 4
  The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" (score of 0) and "worst pain" (score of 100 [100-mm scale]).
Time to advance to regular diet | Up to post-operative day 4
  Time to advance to regular diet through discharge
Time to first ambulation | Up to post-operative day 4
  Time to first ambulation
Return on bowel function | Up to post-operative day 4
  Return on bowel function (pass gas or bowel movement)
Edinburgh Depression scale at hospital discharge (about post-operative day 5) | At hospital discharge (about post-operative day 5)
  The 10-item Edinburgh Depression Scale (EDS) measures depressive symptoms. It includes three sub-scales: anhedonia, anxiety and depression. Possible total scores range from 0 to 30, with higher scores indicating more depressive symptoms and a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zaretsky, MD, Principal Investigator — Children's Hospital Colorado - Colorado Fetal Care Center
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No